CLINICAL TRIAL: NCT05770427
Title: Can We Still Make the Connection? Evaluating an Online Parenting Intervention in a Community-Based Sample of Parents of Infants and Young Children
Brief Title: Evaluating an Online Parenting Intervention in a Community-Based Sample of Parents
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in study design (see NCT05770414 for current and active trial).
Sponsor: University of Ottawa (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H-02-23-8888-2
Record Dates: First submitted 2023-02-21; First posted 2023-03-15 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Parent-Child Relations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental)
  Interventions: Behavioral: Make the Connection® Online Program

INTERVENTIONS:
Behavioral: Make the Connection® Online Program — Make the Connection® (MTC) is an evidence-based parenting program offered by Strong Minds Strong Kids, Psychology Canada. Recently, the MTC program has been adapted to an online platform to help increase scalability and accessibility across Canada. The online modality is self-administered by parents and consist of 8 weekly, 15-minute modules.
  MTC is an attachment-focused, evidence-informed, parent training program that is designed to support the development of positive parent-child relationships by teaching parents to understand their infant's cues. The overarching goal of the program is to enhance parental attitudes and cognitions towards their infants, which have been shown to be associated with sensitive parenting behaviour, and in turn, secure child attachment. Ultimately, by improving parenting skills and attitudes, the program seeks to support secure infant attachment.

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of the online modality of the Make the Connection (MTC) program in a community-based sample of parents not at-risk for parenting difficulties. The main questions it aims to answer are:

* Does the MTC online program result in improvements in parent-child bond, parent self-efficacy, parental stress, and parental depression among parents who are not at-risk for parent-child relationship difficulties?
* What are some of the barriers, facilitators, perceived benefits and risks to participating in the MTC online program from the perspective of parents?

Participants will be asked to complete a pre-intervention questionnaire, will be invited to complete the 8-week MTC online program consisting of a weekly 15-minute module, and will lastly be asked to complete a post-intervention questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* parents with children between the ages of 0-3 years old
* parents are primarily responsible for the children

Exclusion Criteria:

* parents are at-risk for parent-child relationship difficulties (i.e., endorse two of the following criteria: being a first-time caregiver, socially isolated, low education, caregiving alone, lack of confidence or self-efficacy, at risk for poor infant sensitivity, or at-risk for depression)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-06 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Parent-child bond will be measured using the Maternal Postnatal Attachment Scale (MPAS) | Change from pre-intervention scores at baseline and post-intervention scores at week 8
  The MPAS is a 19-item questionnaire that assesses parents' relational attitudes towards their infant. There are three main subscales derived from the measure: Quality of Attachment, Pleasure in Interaction, and Absence of Hostility. The MPAS has shown strong psychometric properties for use in community samples and can be used with mothers and fathers.

SECONDARY OUTCOMES:
Parent self-efficacy will be measured using the Parent Sense of Competence Questionnaire (PSOC) | Change from pre-intervention scores at baseline and post-intervention scores at week 8
  The PSOC has 14-items and measures a parent's experiences in their role as a parent. There are three substances including Interest, Efficacy, and Satisfaction. The questionnaire has been widely used to assess parenting attitudes and has adequate psychometric properties.
Parental stress will be measured using the Parenting Stress Scale (PSS) | Change from pre-intervention scores at baseline and post-intervention scores at week 8
Parental depression will be measured using the Centre for Epidemiological Studies Depression Scale (CES-D) | Change from pre-intervention scores at baseline and post-intervention scores at week 8

CONTACTS AND LOCATIONS:
Locations (1):
- University of Ottawa, Ottawa, Ontario, Canada